CLINICAL TRIAL: NCT00883896
Title: RANDOMIZED, PARALLEL, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ILV-094 ADMINISTERED SUBCUTANEOUSLY TO SUBJECT WITH RHEUMATOID ARTHRITIS.
Brief Title: Study To Evaluate The Safety And Efficacy Of ILV-094 In Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3199K1-2001; B1981001 (Other: Alias Study Number); 2008-006936-37 (EudraCT Number)
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; ACR; Methotrexate; Interleukin-22
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fezakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Placebo Comparator): Part 1: Placebo
  Interventions: Other: Placebo
- Arm 2 (Experimental): Part 1: 100 mg ILV-094 SC Q4W
  Interventions: Drug: ILV-094
- Arm 3 (Experimental): Part 1: 100 mg ILV-094 SC Q2W
  Interventions: Drug: ILV-094
- Arm 4 (Placebo Comparator)
  Interventions: Other: Placebo
- Arm 5 (Experimental): Part 2: 200 mg ILV-094 SC Q2W
  Interventions: Drug: ILV-094

INTERVENTIONS:
Other: Placebo — Part 1: Placebo SC administration every 2 weeks X 10 weeks.
  Arms: Arm 1
Drug: ILV-094 — Part 1: ILV-094 100 mg SC every 4 weeks (alternating ILV-094 100 mg and placebo every 2 weeks) X 10 weeks.
  Arms: Arm 2
Drug: ILV-094 — Part 1: ILV-094 100 mg SC every 2 weeks X 10 weeks.
  Arms: Arm 3
Other: Placebo — Part 2: Placebo SC administration every 2 weeks X 10 weeks
  Arms: Arm 4
Drug: ILV-094 — Part 2: ILV-094 200 mg SC every 2 weeks X 10 weeks
  Arms: Arm 5

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of different dose regimens of ILV-094 compared with placebo, administered subcutaneously to subjects with active rheumatoid arthritis who are taking methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Meets the American College of Rheumatology (ACR) 1987 revised criteria for classification of Rheumatoid Arthritis (RA) for at least 6 months prior to screening
* Active RA at the time of screening and baseline consisting of >= 5 swollen and >= 5 tender joints (28-joint count) and at least 1 of the following at screening: C-reactive protein >= 10 mg/L or Erythrocyte Sedimentation Rate >= 28 mm/h
* Must be receiving methotrexate for at least 12 weeks, with a stable route and dose (up to 25 mg weekly) for at least 8 weeks prior to the baseline visit.

Exclusion Criteria:

* Subjects with other rheumatic diseases
* Cancer or history of cancer (other than cutaneous basal cell carcinoma and squamous cell carcinoma or in situ cervical cancer)
* Any prior use of B cell-depleting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2011-02-18 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (13):
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Center, Palm Harbor, Florida
  - Clinical Research Advantage, Inc., Sarasota, Florida
  - The Arthritis Specialty Centre, Sarasota, Florida
  - Diagnostic Rheumatology and Research PC, Indianapolis, Indiana
  - Clayton Medical Research, St Louis, Missouri
  - Deaconess Hospital, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, West Reading, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Arthritis Care and Diagnostic Center, Dallas, Texas
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas
- Belgium (5):
  - AZ Jan Palfijn, Antwerp
  - Cliniques Universitaires St Luc Avenue Hippocrate 10 UCL, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Reuma Instituut, Hasselt
  - Chu Liege Sart Tilman B 35, Liège
- Colombia (4):
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogota, Cundinamarca
  - Medicity S.A.S, Bucaramanga, Santander Department
  - Servimed EU, Bucaramanga, Santander Department
- Croatia (2):
  - University Hospital Centre Rijeka, Rijeka
  - University Hospital Center Zagreb, Zagreb
- Klinikum Innenstadt der Ludwig-Maximillians-Universität, München, Germany
- Hungary (4):
  - Budai Irgalmasrendi Hospital, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Josa Andras Oktatokorhaz Egeszsegugyi Szolgaltato Nonprofit Kft., Nyíregyháza
  - Markusovszky Hospital, Szombathely
- Japan (8):
  - National Hospital Organization Shimoshizu National Hospital, Yotsukaidou, Chiba
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Medical Corporation Wakoukai Kurashiki Kousai Hospital, Kurashiki, Okayama-ken
  - Institute of Rheumatology, Tokyo Women's Medical University Hospital, Shinjyuku-ku, Tokyo
  - Inoue Hospital, Gunma
  - Matsubara Clinic, Hyōgo
  - Matsubara Mayflower Hospital, Hyōgo
- Centro de Estudio de Investigacion Basica y Clinica S.C, Jalisco, Guadalajara, Mexico
- AMC, Amsterdam, North Holland, Netherlands
- Romania (6):
  - Centrul Medical Terra Med, Cluj-Napoca, Cluj
  - SC Duo Medical SRL, Bucharest
  - Spitalul Clinic Sf. Maria, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Centrul de Boli Reumatismale Dr. I. Stoia, Bucharest
  - Spitalul Clinic Judetean de Urgenta Tg Mures, Târgu Mureş
- Russia (7):
  - Institute of Rheumatology of Russian academy of Medical Scie, Moscow
  - City Clinical Hospital # 1 n.a. Pirogov, Moscow
  - State Educational Institution of Additional Professional Education, Saint Petersburg
  - State Health care institution of Leningrad Regional Clinical Hospital, Saint Petersburg
  - State education institution of higher vocational education Smolensk State Medical Academy Roszdrav, Smolensk
  - State Healthcare Institution Yaroslavl Regional Clinical Hospital, Yaroslavl
  - Municipal Institution City Clinical Hospital #40, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=3199K1-2001

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to ILV-094 subcutaneous injection at Day 1 and then every 2 weeks up to Week 10. Participants were followed up to 12 weeks after last study drug administration.
- ILV-094 100 mg Every 4 Weeks: Participants received ILV-094 100 milligram (mg) subcutaneous injection at Day 1 and then every 4 weeks up to Week 10. Participants were followed up to 12 weeks after last study drug administration.
- ILV-094 100 mg Every 2 Weeks: Participants received ILV-094 100 mg subcutaneous injection at Day 1 and then every 2 weeks up to Week 10. Participants were followed up to 12 weeks after last study drug administration.
- ILV-094 200 mg Every 2 Weeks: Participants received ILV-094 200 mg subcutaneous injection at Day 1 and then every 2 weeks up to Week 10. Participants were followed up to 12 weeks after last study drug administration.
Period: Overall Study
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Started | 66 | 39 | 42 | 48
Completed | 60 | 39 | 41 | 41
Not Completed | 6 | 0 | 1 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 5 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks | Total
Number analyzed (Participants) | 66 | 39 | 42 | 48 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.91 (11.01) | 59.95 (10.30) | 55.14 (10.80) | 54.90 (11.11) | 56.64 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 34 | 31 | 38 | 156
  Male | 13 | 5 | 11 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20 Percent (ACR20) Response at Week 12
Description: ACR20 response: greater than or equal to (>=) 20 percent improvement in tender joint count; >=20 percent improvement in swollen joint count; and >=20 percent improvement in 3 of 5 remaining ACR core measures: participant's global assessment of disease activity (score: 0 [very well] to 10 [worst]); participant's assessment of pain (score: 0 [very well] to 100 [extremely bad]); physician global assessment of disease activity (score: 0 [very well] to 10 [worst]); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]) (score: 0 [no difficulty] to 3 [unable to do]); and C-reactive protein (CRP).
Time Frame: Week 12
Population: mITT population included all randomized participants who received at least 1 dose of study drug. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Percentage of participants | 50.0 [37.4 to 62.6] | 43.6 [27.8 to 60.4] | 38.1 [23.6 to 54.4] | 50.0 [35.2 to 64.8]
Statistical Analysis 1: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; P-value was assessed from 2-sided Cochran-Mantel-Haenszel (CMH) test stratified by anti-tumor necrosis factor (anti-TNF) prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.558, Cochran-Mantel-Haenszel; Percent Difference = -5.9, 95% CI 2-sided [-25.0 to 13.3]
Statistical Analysis 2: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.251, Cochran-Mantel-Haenszel; Percent Difference = -11.4, 95% CI 2-sided [-30.1 to 7.3]
Statistical Analysis 3: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.707, Cochran-Mantel-Haenszel; Percent Difference = -3.7, 95% CI 2-sided [-21.7 to 14.4]

2. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20 Percent (ACR20) Response at Week 2, 4, 6, 8 and 10
Description: ACR20 response: >=20 percent improvement in tender joint count; >=20 percent improvement in swollen joint count; and >=20 percent improvement in 3 of 5 remaining ACR core measures: participant's global assessment of disease activity (score: 0 [very well] to 10 [worst]); participant's assessment of pain (score: 0 [very well] to 100 [extremely bad]); physician global assessment of disease activity (score: 0 [very well] to 10 [worst]); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]) (score: 0 [no difficulty] to 3 [unable to do]); and C-reactive protein (CRP).
Time Frame: Week 2, 4, 6, 8, 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug. LOCF method was used to impute missing values.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Percentage of participants
  Week 2 | 18.2 [9.8 to 29.6] | 17.9 [7.5 to 33.5] | 14.3 [5.4 to 28.5] | 14.6 [6.1 to 27.8]
  Week 4 | 24.2 [14.5 to 36.4] | 33.3 [19.1 to 50.2] | 21.4 [10.3 to 36.8] | 27.1 [15.3 to 41.8]
  Week 6 | 33.3 [22.2 to 46.0] | 46.2 [30.1 to 62.8] | 23.8 [12.1 to 39.5] | 39.6 [25.8 to 54.7]
  Week 8 | 31.8 [20.9 to 44.4] | 48.7 [32.4 to 65.2] | 33.3 [19.6 to 49.5] | 35.4 [22.2 to 50.5]
  Week 10 | 42.4 [30.3 to 55.2] | 56.4 [39.6 to 72.2] | 42.9 [27.7 to 59.0] | 31.3 [18.7 to 46.3]
Statistical Analysis 1: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 2: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.991, Cochran-Mantel-Haenszel; Percent Difference = -0.1, 95% CI 2-sided [-14.8 to 14.7]
Statistical Analysis 2: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.518, Cochran-Mantel-Haenszel; Percent Difference = -4.8, 95% CI 2-sided [-18.4 to 8.8]
Statistical Analysis 3: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.630, Cochran-Mantel-Haenszel; Perecent Difference = 0.781, 95% CI 2-sided [-16.9 to 9.8]
Statistical Analysis 4: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 4: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.295, Cochran-Mantel-Haenszel; Percent Difference = 9.4, 95% CI 2-sided [-8.3 to 27.0]
Statistical Analysis 5: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.686, Cochran-Mantel-Haenszel; Perecent Difference = -3.4, 95% CI 2-sided [-19.3 to 12.5]
Statistical Analysis 6: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.772, Cochran-Mantel-Haenszel; Percent Difference = 2.5, 95% CI 2-sided [-13.2 to 18.2]
Statistical Analysis 7: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 6: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.201, Cochran-Mantel-Haenszel; Percent Difference = 12.8, 95% CI 2-sided [-6.5 to 32.0]
Statistical Analysis 8: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.256, Cochran-Mantel-Haenszel; Percent Difference = -10.4, 95% CI 2-sided [-27.3 to 6.5]
Statistical Analysis 9: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.519, Cochran-Mantel-Haenszel; Percent Difference = 6.1, 95% CI 2-sided [-11.4 to 23.5]
Statistical Analysis 10: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 8: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.094, Cochran-Mantel-Haenszel; Percent Difference = 16.7, 95% CI 2-sided [-1.9 to 35.2]
Statistical Analysis 11: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.760, Cochran-Mantel-Haenszel; Percent Difference = 2.8, 95% CI 2-sided [-14.4 to 20.1]
Statistical Analysis 12: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.950, Cochran-Mantel-Haenszel; Percent Difference = 0.6, 95% CI 2-sided [-16.8 to 18.0]
Statistical Analysis 13: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 10: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.185, Cochran-Mantel-Haenszel; Percent Difference = 13.6, 95% CI 2-sided [-5.9 to 33.0]
Statistical Analysis 14: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.982, Cochran-Mantel-Haenszel; Percent Difference = 0.2, 95% CI 2-sided [-18.8 to 19.3]
Statistical Analysis 15: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.223, Cochran-Mantel-Haenszel; Percent Difference = -11.6, 95% CI 2-sided [-29.0 to 5.8]

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50 Percent (ACR50) Response at Week 2, 4, 6, 8, 10 and 12
Description: ACR50 response: >=50 percent improvement in tender joint count; >=50 percent improvement in swollen joint count; and 50 improvement in 3 of 5 remaining ACR core measures: participant's global assessment of disease activity (score: 0 [very well] to 10 [worst]); participant's assessment of pain (score: 0 [very well] to 100 [extremely bad]); physician global assessment of disease activity (score: 0 [very well] to 10 [worst]); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]) (score: 0 [no difficulty] to 3 [unable to do]); and C-reactive protein (CRP).
Time Frame: Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Percentage of participants
  Week 2 | 3.0 [0.4 to 10.5] | 2.6 [0.1 to 13.5] | 9.5 [2.7 to 22.6] | 0.0 [0.0 to 7.4]
  Week 4 | 6.1 [1.7 to 14.8] | 7.7 [1.6 to 20.9] | 7.1 [1.5 to 19.5] | 4.2 [0.5 to 14.3]
  Week 6 | 9.1 [3.4 to 18.7] | 7.7 [1.6 to 20.9] | 14.3 [5.4 to 28.5] | 12.5 [4.7 to 25.2]
  Week 8 | 7.6 [2.5 to 16.8] | 12.8 [4.3 to 27.4] | 4.8 [0.6 to 16.2] | 14.6 [6.1 to 27.8]
  Week 10 | 18.2 [9.8 to 29.6] | 17.9 [7.5 to 33.5] | 9.5 [2.7 to 22.6] | 18.8 [8.9 to 32.6]
  Week 12 | 15.2 [7.5 to 26.1] | 23.1 [11.1 to 39.3] | 14.3 [5.4 to 28.5] | 14.6 [6.1 to 27.8]
Statistical Analysis 1: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.885, Cochran-Mantel-Haenszel; Percent Difference = -0.5, 95% CI 2-sided [-6.8 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.180, Cochran-Mantel-Haenszel; Percent Difference = 6.1, 95% CI 2-sided [-3.4 to 15.6]
Statistical Analysis 3: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.277, Cochran-Mantel-Haenszel; Percent Difference = -2.7, 95% CI 2-sided [-6.5 to 1.1]
Statistical Analysis 4: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.740, Cochran-Mantel-Haenszel; Percent Difference = 1.7, 95% CI 2-sided [-7.9 to 11.3]
Statistical Analysis 5: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.934, Cochran-Mantel-Haenszel; Percent Difference = 0.4, 95% CI 2-sided [-9.3 to 10.1]
Statistical Analysis 6: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.876, Cochran-Mantel-Haenszel; Percent Difference = -0.6, 95% CI 2-sided [-7.7 to 6.4]
Statistical Analysis 7: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.842, Cochran-Mantel-Haenszel; Percent Difference = -1.1, 95% CI 2-sided [-11.4 to 9.2]
Statistical Analysis 8: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.509, Cochran-Mantel-Haenszel; Percent Difference = 4.1, 95% CI 2-sided [-8.1 to 16.3]
Statistical Analysis 9: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.504, Cochran-Mantel-Haenszel; Percent Difference = 4.0, 95% CI 2-sided [-7.0 to 15.0]
Statistical Analysis 10: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.373, Cochran-Mantel-Haenszel; Percent Difference = 5.4, 95% CI 2-sided [-6.3 to 17.0]
Statistical Analysis 11: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.499, Cochran-Mantel-Haenszel; Percent Difference = -3.4, 95% CI 2-sided [-12.0 to 5.2]
Statistical Analysis 12: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.244, Cochran-Mantel-Haenszel; Percent Difference = 7.0, 95% CI 2-sided [-4.2 to 18.3]
Statistical Analysis 13: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.979, Cochran-Mantel-Haenszel; Percent Difference = -0.2, 95% CI 2-sided [-15.0 to 14.6]
Statistical Analysis 14: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.166, Cochran-Mantel-Haenszel; Percent Difference = -9.8, 95% CI 2-sided [-21.8 to 2.2]
Statistical Analysis 15: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.947, Cochran-Mantel-Haenszel; Percent Difference = 0.5, 95% CI 2-sided [-13.2 to 14.2]
Statistical Analysis 16: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 12: P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.286, Cochran-Mantel-Haenszel; Percent Difference = 8.3, 95% CI 2-sided [-7.1 to 23.8]
Statistical Analysis 17: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.822, Cochran-Mantel-Haenszel; Percent Difference = -1.6, 95% CI 2-sided [-15.0 to 11.8]
Statistical Analysis 18: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.986, Cochran-Mantel-Haenszel; Percent Difference = -0.1, 95% CI 2-sided [-12.3 to 12.1]

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70 Percent (ACR70) Response at Week 2, 4, 6, 8, 10 and 12
Description: ACR70 response:>=70 percent improvement in tender joint count; >=70 percent improvement in swollen joint count; and 70 percent improvement in 3 of 5 remaining ACR core measures: participant's global assessment of disease activity (score: 0 [very well] to 10 [worst]); participant's assessment of pain (score: 0 [very well] to 100 [extremely bad]); physician global assessment of disease activity (score: 0 [very well] to 10 [worst]); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]) (score: 0 [no difficulty] to 3 [unable to do]); and C-reactive protein (CRP).
Time Frame: Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Percentage of participants
  Week 2 | 0.0 [0.0 to 5.4] | 2.6 [0.1 to 13.5] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 7.4]
  Week 4 | 1.5 [0.0 to 8.2] | 2.6 [0.1 to 13.5] | 7.1 [1.5 to 19.5] | 0.0 [0.0 to 7.4]
  Week 6 | 0.0 [0.0 to 5.4] | 2.6 [0.1 to 13.5] | 2.4 [0.1 to 12.6] | 2.1 [0.1 to 11.1]
  Week 8 | 0.0 [0.0 to 5.4] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 8.4] | 4.2 [0.5 to 14.3]
  Week 10 | 0.0 [0.0 to 5.4] | 5.1 [0.6 to 17.3] | 2.4 [0.1 to 12.6] | 2.1 [0.1 to 11.1]
  Week 12 | 4.5 [0.9 to 12.7] | 5.1 [0.6 to 17.3] | 4.8 [0.6 to 16.2] | 2.1 [0.1 to 11.1]
Statistical Analysis 1: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.205, Cochran-Mantel-Haenszel; Percent Difference = 2.5, 95% CI 2-sided [-2.3 to 7.4]
Statistical Analysis 2: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; Week 2:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.188, Cochran-Mantel-Haenszel; Percent Difference = 2.5, 95% CI 2-sided [-2.3 to 7.3]
Statistical Analysis 3: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; Week 2: Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 4: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 4:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.699, Cochran-Mantel-Haenszel; Percent Difference = 1.1, 95% CI 2-sided [-4.5 to 6.6]
Statistical Analysis 5: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.155, Cochran-Mantel-Haenszel; Percent Difference = 5.4, 95% CI 2-sided [-3.0 to 13.8]
Statistical Analysis 6: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.546, Cochran-Mantel-Haenszel; Percent Difference = -1.0, 95% CI 2-sided [-2.9 to 0.9]
Statistical Analysis 7: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 6:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.205, Cochran-Mantel-Haenszel; Percent Difference = 2.5, 95% CI 2-sided [-2.3 to 7.4]
Statistical Analysis 8: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.269, Cochran-Mantel-Haenszel; Percent Difference = 2.2, 95% CI 2-sided [-1.8 to 6.1]
Statistical Analysis 9: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.723, Cochran-Mantel-Haenszel; Percent Difference = 2.0, 95% CI 2-sided [-1.6 to 5.6]
Statistical Analysis 10: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.205, Cochran-Mantel-Haenszel; Percent Difference = 2.5, 95% CI 2-sided [-2.3 to 7.4]
Statistical Analysis 11: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; Week 8: Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the cochran method; Test type: Superiority or Other; Percent Difference = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 12: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; Week 8:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.125, Cochran-Mantel-Haenszel; Percent Difference = 4.0, 95% CI 2-sided [-1.3 to 9.4]
Statistical Analysis 13: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 10:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.071, Cochran-Mantel-Haenszel; Percent Difference = 5.0, 95% CI 2-sided [-1.7 to 11.8]
Statistical Analysis 14: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel; Percent Difference = 2.0, 95% CI 2-sided [-1.2 to 5.1]
Statistical Analysis 15: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.280, Cochran-Mantel-Haenszel; Percent Difference = 2.0, 95% CI 2-sided [-1.6 to 5.6]
Statistical Analysis 16: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 12:P-value was assessed from 2-sided CMH test stratified by anti-TNF prior use and geographic region of the site. Treatment group differences and the corresponding confidence intervals adjusted for stratification were calculated using the Cochran method; Test type: Superiority or Other; p = 0.892, Cochran-Mantel-Haenszel; Percent Difference = 0.6, 95% CI 2-sided [-7.6 to 8.8]
Statistical Analysis 17: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.903, Cochran-Mantel-Haenszel; Percent Difference = -0.5, 95% CI 2-sided [-8.3 to 7.2]
Statistical Analysis 18: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.625, Cochran-Mantel-Haenszel; Percent Difference = -1.7, 95% CI 2-sided [-7.2 to 3.8]

5. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28) Using C-Reactive Protein (CRP)
Description: DAS28 (CRP) was calculated from number of swollen joints and tender joints using the 28 joints count; CRP (milligram/Liter [mg/L]); and general health visual analog scale (VAS) score (participant rated scale with scores ranging from 0mm [very well] to 100mm [extremely bad]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28 (CRP) less than or equal to (<=) 3.2 implied low disease activity, greater than (>) 3.2 to 5.1 implied moderate to high disease activity, and less than (<) 2.6 implied remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: mITT population included all randomized participants who received at least 1 dose of study drug. LOCF method was used to impute missing values. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline: number analyzed (Participants) | 65 | 39 | 42 | 48
  Baseline | 5.6 (0.8) | 5.5 (0.9) | 5.3 (0.8) | 5.5 (0.8)
  Week 2 | 5.1 (1.0) | 5.1 (1.1) | 4.9 (1.4) | 5.2 (1.0)
  Week 4 | 4.9 (1.1) | 4.8 (0.9) | 4.6 (1.4) | 5.0 (1.1)
  Week 6 | 4.7 (1.2) | 4.4 (1.2) | 4.6 (1.2) | 4.6 (1.2)
  Week 8 | 4.6 (1.3) | 4.4 (1.1) | 4.4 (1.2) | 4.4 (1.3)
  Week 10 | 4.5 (1.3) | 4.2 (1.2) | 4.4 (1.2) | 4.5 (1.3)
  Week 12 | 4.4 (1.3) | 4.2 (1.4) | 4.3 (1.3) | 4.4 (1.3)

6. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28) Using Erythrocyte Sedimentation Rate (ESR)
Description: DAS28 (ESR) was calculated from the number of swollen joints and tender joints using the 28 joints count; ESR (millimeters per hour [mm/hour]); and general health VAS score (participant rated scale with scores ranging from 0 [very well] to 100 [extremely bad]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28 (ESR) <=3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity, and <2.6 implied remission.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: mITT population included all randomized participants who received at least 1 or even partial dose of study drug. LOCF method was used to impute missing values. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline: number analyzed (Participants) | 65 | 39 | 42 | 48
  Baseline | 6.4 (0.7) | 6.4 (0.8) | 6.2 (0.7) | 6.3 (0.8)
  Week 2 | 5.8 (1.1) | 5.9 (1.1) | 5.6 (1.4) | 5.9 (0.8)
  Week 4 | 5.5 (1.3) | 5.6 (0.9) | 5.3 (1.3) | 5.7 (0.9)
  Week 6 | 5.4 (1.3) | 5.2 (1.1) | 5.3 (1.2) | 5.2 (1.2)
  Week 8 | 5.3 (1.3) | 5.2 (1.1) | 5.0 (1.3) | 5.1 (1.2)
  Week 10 | 5.2 (1.4) | 5.0 (1.2) | 5.0 (1.3) | 5.1 (1.3)
  Week 12 | 5.1 (1.3) | 5.0 (1.4) | 5.0 (1.3) | 5.1 (1.3)

7. Secondary Outcome: Tender Joints Counts (TJC)
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Tender joints
  Baseline | 13.4 (5.2) | 13.2 (6.3) | 12.3 (5.9) | 14.4 (5.9)
  Week 2 | 11.1 (6.0) | 10.9 (7.1) | 10.8 (7.8) | 12.5 (6.4)
  Week 4 | 10.4 (6.6) | 9.5 (7.1) | 9.5 (6.7) | 11.2 (6.5)
  Week 6 | 9.5 (7.1) | 8.1 (7.5) | 9.2 (7.8) | 9.3 (6.4)
  Week 8 | 9.2 (7.2) | 7.8 (7.2) | 7.9 (7.2) | 9.3 (6.6)
  Week 10 | 8.4 (7.0) | 7.2 (6.9) | 8.0 (7.1) | 9.5 (7.0)
  Week 12 | 7.7 (6.4) | 7.4 (8.0) | 7.8 (7.7) | 9.2 (7.0)

8. Secondary Outcome: Swollen Joints Count (SJC)
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Swollen joints
  Baseline | 10.2 (3.8) | 10.0 (4.6) | 9.4 (4.6) | 10.0 (4.1)
  Week 2 | 8.2 (5.0) | 8.4 (5.2) | 6.9 (5.2) | 8.0 (4.7)
  Week 4 | 7.0 (4.9) | 6.8 (5.1) | 5.8 (5.0) | 7.0 (5.0)
  Week 6 | 6.6 (5.3) | 5.7 (5.4) | 6.0 (5.8) | 5.9 (5.1)
  Week 8 | 6.4 (5.4) | 6.0 (6.0) | 5.0 (4.9) | 5.6 (5.2)
  Week 10 | 5.9 (5.8) | 5.4 (5.5) | 5.2 (5.2) | 5.9 (5.8)
  Week 12 | 5.5 (5.6) | 5.6 (5.9) | 5.0 (5.3) | 5.5 (5.9)

9. Secondary Outcome: Physician Global Assessment of Disease Activity
Description: Physician global assessment of disease activity was measured on an 11-point scale, ranging from 0 to 10, where 0 = no disease activity and 10 = extreme disease activity.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline | 6.2 (1.6) | 6.3 (1.5) | 6.0 (1.7) | 6.0 (1.6)
  Week 2 | 5.4 (1.9) | 5.2 (1.8) | 5.1 (2.1) | 5.1 (1.7)
  Week 4 | 4.7 (1.9) | 4.9 (1.8) | 4.6 (2.2) | 4.9 (1.9)
  Week 6 | 4.4 (1.8) | 4.5 (1.9) | 4.3 (1.8) | 4.3 (2.0)
  Week 8 | 4.5 (2.1) | 3.9 (1.6) | 3.9 (1.9) | 4.1 (2.0)
  Week 10 | 4.2 (2.3) | 3.6 (1.7) | 3.9 (1.9) | 4.2 (2.3)
  Week 12 | 4.0 (2.2) | 3.7 (2.1) | 3.6 (1.9) | 3.9 (2.1)

10. Secondary Outcome: Participant Global Assessment of Disease Activity
Description: Participants answered: "considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a scale ranging from 0 to 10, where 0 = no disease activity and 10 = extreme disease activity.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline | 6.2 (1.8) | 6.0 (1.8) | 6.3 (1.7) | 5.9 (2.1)
  Week 2 | 5.5 (2.3) | 5.5 (2.1) | 5.6 (2.4) | 5.7 (2.2)
  Week 4 | 5.2 (2.1) | 5.0 (2.2) | 5.6 (2.2) | 5.5 (2.0)
  Week 6 | 5.0 (2.0) | 4.7 (2.2) | 5.4 (1.8) | 5.1 (2.1)
  Week 8 | 5.1 (2.1) | 4.6 (2.3) | 5.5 (1.9) | 4.8 (2.0)
  Week 10 | 5.0 (2.3) | 4.0 (2.4) | 5.2 (2.1) | 5.0 (2.2)
  Week 12 | 4.7 (2.1) | 4.5 (2.4) | 5.0 (2.0) | 4.8 (2.2)

11. Secondary Outcome: Pain Visual Analog Scale (VAS)
Description: Participants assessed the amount of pain currently experienced by them on a 100 millimeter (mm) VAS ranging from 0= no pain to 100= severe pain.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Millimeter
  Baseline | 58.0 (21.2) | 56.0 (19.1) | 56.6 (18.7) | 56.5 (23.6)
  Week 2 | 49.8 (23.5) | 48.3 (24.0) | 51.7 (23.7) | 52.3 (21.5)
  Week 4 | 46.8 (23.7) | 45.9 (23.9) | 54.7 (22.0) | 52.6 (20.7)
  Week 6 | 48.8 (23.6) | 45.2 (23.5) | 48.8 (18.9) | 46.7 (21.7)
  Week 8 | 47.3 (24.4) | 38.9 (23.5) | 49.0 (22.8) | 44.1 (21.2)
  Week 10 | 45.2 (26.1) | 37.7 (24.6) | 46.2 (24.0) | 44.7 (23.5)
  Week 12 | 44.0 (25.0) | 39.9 (23.9) | 44.9 (22.4) | 42.6 (19.9)

12. Secondary Outcome: General Health Visual Analog Scale (VAS)
Description: General health VAS is a 100 mm line marked by the participant. Participants were asked, "In general how would you rate your health currently concerning the arthritis?" Scores ranged from 0 mm = very well to 100 mm = extremely bad.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12
Population: mITT population included all randomized participants who received at least 1 dose of study drug. LOCF method was used to impute missing values. Here 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Millimeter
  Baseline: number analyzed (Participants) | 65 | 39 | 42 | 48
  Baseline | 60.8 (18.4) | 59.2 (21.2) | 61.0 (16.4) | 57.7 (20.7)
  Week 2 | 54.1 (22.4) | 52.5 (23.0) | 53.0 (23.7) | 54.8 (19.8)
  Week 4 | 48.8 (23.0) | 48.2 (22.9) | 54.3 (23.1) | 52.9 (20.2)
  Week 6 | 50.7 (22.0) | 42.4 (21.9) | 52.5 (19.4) | 48.8 (21.9)
  Week 8 | 47.5 (24.1) | 40.4 (23.8) | 50.3 (22.2) | 45.4 (21.5)
  Week 10 | 48.4 (25.7) | 38.9 (22.2) | 46.9 (24.0) | 45.7 (23.3)
  Week 12 | 47.6 (25.4) | 40.6 (23.0) | 47.4 (22.0) | 43.2 (21.4)

13. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: Health assessment questionnaire-disability index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to perform activity. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Week 4, 2, 6, 8, 10, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline | 1.4 (0.7) | 1.3 (0.7) | 1.3 (0.6) | 1.3 (0.7)
  Week 2 | 1.3 (0.7) | 1.3 (0.7) | 1.2 (0.7) | 1.3 (0.6)
  Week 4 | 1.3 (0.7) | 1.1 (0.6) | 1.3 (0.7) | 1.2 (0.7)
  Week 6 | 1.2 (0.7) | 1.1 (0.7) | 1.2 (0.6) | 1.2 (0.7)
  Week 8 | 1.2 (0.6) | 1.1 (0.7) | 1.2 (0.7) | 1.1 (0.7)
  Week 10 | 1.2 (0.7) | 1.1 (0.7) | 1.2 (0.7) | 1.1 (0.7)
  Week 12 | 1.2 (0.7) | 1.1 (0.7) | 1.1 (0.7) | 1.1 (0.7)

14. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey consisting of 36 items summarized into 8 multi-item scales evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality and mental health. Two summary scores, the physical component summary (PCS) and the mental component summary (MCS) derived are derived by aggregating the 8 aspects. The score for each aspect and physical and mental component summary are scaled 0-100 where, higher score indicating highest level of functioning.
Time Frame: Baseline, Week 4, 8, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline: PCS: number analyzed (Participants) | 65 | 39 | 42 | 48
  Baseline: PCS | 33.8 (7.8) | 34.9 (5.8) | 34.8 (6.6) | 34.4 (8.3)
  Baseline: MCS: number analyzed (Participants) | 65 | 39 | 42 | 48
  Baseline: MCS | 40.5 (12.3) | 42.0 (12.0) | 41.2 (11.0) | 41.1 (13.0)
  Week 4: PCS | 36.0 (8.2) | 36.9 (8.5) | 36.0 (8.6) | 36.5 (7.7)
  Week 4: MCS | 42.7 (12.4) | 43.0 (13.0) | 41.0 (12.2) | 40.3 (12.4)
  Week 8: PCS | 35.8 (7.5) | 37.3 (8.5) | 36.6 (7.1) | 36.9 (8.1)
  Week 8: MCS | 44.5 (11.3) | 44.8 (12.0) | 43.1 (11.9) | 42.9 (11.3)
  Week 12: PCS | 36.7 (7.7) | 37.6 (8.6) | 36.3 (8.7) | 37.1 (9.4)
  Week 12: MCS | 43.2 (11.8) | 44.2 (11.7) | 44.2 (12.6) | 44.5 (9.8)

15. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-fatigue is a 13-item questionnaire. Participants score each item on a 5-point scale ranging from 0 (not at all) to 4 (very much). The scoring algorithm is such that the item responses are reversed in score (except for 2 items, "I have energy" and "I am able to do my usual activities"), in order to reflect higher scores as less fatigue. The sum of all responses resulted in the FACIT-fatigue total score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Week 4, 8, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Units on a scale
  Baseline | 29.1 (10.9) | 30.9 (10.9) | 30.6 (9.4) | 29.2 (11.7)
  Week 4 | 31.7 (10.7) | 33.6 (11.3) | 32.6 (9.8) | 30.7 (10.6)
  Week 8 | 32.7 (10.8) | 33.7 (10.4) | 32.1 (9.9) | 32.3 (10.7)
  Week 12 | 33.3 (9.4) | 34.3 (9.5) | 32.4 (9.5) | 33.2 (10.9)

16. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: DAS28-based EULAR response criteria was used to measure individual response as none, good and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1.
Time Frame: Week 2, 4, 6, 8, 10, 12
Population: mITT population included all randomized participants who received at least 1 dose of study drug. LOCF method was used to impute missing values. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Number analyzed (Participants) | 66 | 39 | 42 | 48
Participants
  Week 2: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 2: Good | 3 | 1 | 5 | 0
  Week 2: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 2: Moderate | 15 | 10 | 7 | 9
  Week 2: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 2: None | 47 | 28 | 30 | 39
  Week 4: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 4: Good | 4 | 2 | 6 | 1
  Week 4: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 4: Moderate | 20 | 13 | 9 | 15
  Week 4: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 4: None | 41 | 24 | 27 | 32
  Week 6: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 6: Good | 7 | 4 | 4 | 5
  Week 6: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 6: Moderate | 27 | 20 | 11 | 18
  Week 6: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 6: None | 31 | 15 | 27 | 25
  Week 8: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 8: Good | 8 | 5 | 4 | 8
  Week 8: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 8: Moderate | 29 | 18 | 16 | 19
  Week 8: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 8: None | 28 | 16 | 22 | 21
  Week 10: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 10: Good | 13 | 6 | 6 | 7
  Week 10: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 10: Moderate | 28 | 22 | 15 | 21
  Week 10: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 10: None | 24 | 11 | 21 | 20
  Week 12: Good: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 12: Good | 12 | 11 | 7 | 9
  Week 12: Moderate: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 12: Moderate | 33 | 16 | 18 | 20
  Week 12: None: number analyzed (Participants) | 65 | 39 | 42 | 48
  Week 12: None | 20 | 12 | 17 | 19
Statistical Analysis 1: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 2: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.900, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.522, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.147, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.534, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.206, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.070, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 4: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.936, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.625, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.586, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.685, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.340, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 7]; Test type: Superiority or Other; p = 0.212, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 6: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.455, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.145, Cochran-Mantel-Haenszel
Statistical Analysis 15: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.660, Cochran-Mantel-Haenszel
Statistical Analysis 16: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.050, Cochran-Mantel-Haenszel
Statistical Analysis 17: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.428, Cochran-Mantel-Haenszel
Statistical Analysis 18: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 13]; Test type: Superiority or Other; p = 0.160, Cochran-Mantel-Haenszel
Statistical Analysis 19: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 8: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.757, Cochran-Mantel-Haenszel
Statistical Analysis 20: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.408, Cochran-Mantel-Haenszel
Statistical Analysis 21: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.983, Cochran-Mantel-Haenszel
Statistical Analysis 22: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.374, Cochran-Mantel-Haenszel
Statistical Analysis 23: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.992, Cochran-Mantel-Haenszel
Statistical Analysis 24: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 19]; Test type: Superiority or Other; p = 0.422, Cochran-Mantel-Haenszel
Statistical Analysis 25: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 10: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.743, Cochran-Mantel-Haenszel
Statistical Analysis 26: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.188, Cochran-Mantel-Haenszel
Statistical Analysis 27: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.385, Cochran-Mantel-Haenszel
Statistical Analysis 28: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.148, Cochran-Mantel-Haenszel
Statistical Analysis 29: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.304, Cochran-Mantel-Haenszel
Statistical Analysis 30: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 25]; Test type: Superiority or Other; p = 0.552, Cochran-Mantel-Haenszel
Statistical Analysis 31: Comparison: Placebo vs ILV-094 100 mg Every 4 Weeks; Week 12: P-value was assessed from 2-sided stratified CMH row mean test by anti-TNF prior use and geographic region of the site; Test type: Superiority or Other; p = 0.494, Cochran-Mantel-Haenszel
Statistical Analysis 32: Comparison: Placebo vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.421, Cochran-Mantel-Haenszel
Statistical Analysis 33: Comparison: Placebo vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.418, Cochran-Mantel-Haenszel
Statistical Analysis 34: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 100 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.235, Cochran-Mantel-Haenszel
Statistical Analysis 35: Comparison: ILV-094 100 mg Every 4 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.268, Cochran-Mantel-Haenszel
Statistical Analysis 36: Comparison: ILV-094 100 mg Every 2 Weeks vs ILV-094 200 mg Every 2 Weeks; [analysis description as in outcome 16, analysis 31]; Test type: Superiority or Other; p = 0.957, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | ILV-094 100 mg Every 4 Weeks | ILV-094 100 mg Every 2 Weeks | ILV-094 200 mg Every 2 Weeks
Serious Adverse Events (participants affected / at risk) | 7/66 | 2/39 | 0/42 | 0/48
Other Adverse Events (participants affected / at risk) | 35/66 | 29/39 | 26/42 | 28/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | ILV-094 100 mg Every 4 Weeks (N=39) | ILV-094 100 mg Every 2 Weeks (N=42) | ILV-094 200 mg Every 2 Weeks (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Testicular abscess (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | ILV-094 100 mg Every 4 Weeks (N=39) | ILV-094 100 mg Every 2 Weeks (N=42) | ILV-094 200 mg Every 2 Weeks (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Presbyopia (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Apical granuloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 2 | 2
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 1 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2 | 1
Herpes zoster (Infections and infestations) | 2 | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4 | 4
Oral herpes (Infections and infestations) | 1 | 0 | 3 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 2 | 2 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 2
Blood pressure increased (Investigations) | 2 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 1
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0
Listless (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Calculus prostatic (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema weeping (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Varicose ulceration (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.